CLINICAL TRIAL: NCT03491891
Title: Correlates and Mehcanisms Underlying Very Late Stent Thrombosis After Implantation of New Generation DES in China
Brief Title: Factors Contribute to Very Late Stent Thrombosis After New Generation DES Implantation in China
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: First Affiliated Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: wx19871203
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2018-06

CONDITIONS: Stent Thrombosis
Keywords: Very Late Stent Thrombosis; New generation DES

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — blood samples including serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- derivation cohort: no interventions will be administrated
- validation cohort: no interventions will be administrated

SUMMARY:
The investigators sought to identify and verify the potential correlates and mechanisms of Very Late Stent Thrombosis (VLST) after the implantation of new generation drug eluting steng in China from an analysis of multicenter registries.

DETAILED DESCRIPTION:
This study represents a patient-level pooled analysis of patients undergoing percutaneous coronary intervention with stent implantation for acute coronary syndrome. Multiple aspects including clinical, angiographic, procedural characteristics , intravascular imaging results and blood samples were collected at index PCI and the time of VLST or CAG during follow-up, in order to reveal the potential mechanisms or risk factors that contribute to the development of VLST.

ELIGIBILITY:
Inclusion Criteria:

* Patients>18y,admitted for acute coronary syndrome,successfully underwent PCI with at least one stent, sign informed consent.

Exclusion Criteria:

* Expected lifetime was less than 1 year for any severe disease(such as tumor,severe respiratory failure et al). There is a surgical plan for important organs within 1 year after surgery and anti-platelet drugs should be discontinued. Refusing to sign informed consent.Died prior to discharge. Poor compliance, unable to participate in regular follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients>18y,admitted for acute coronary syndrome,successfully underwent PCI with at least one stent, sign informed consent were included.Patients' expected lifetime was less than 1 year for any severe disease(such as tumor,severe respiratory failure et al),and with a surgical plan for important organs within 1 year after surgery and anti-platelet drugs should be discontinued, refusing to sign informed consent, died prior to discharge, unable to participate in regular follow-up were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 8476 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: yang zheng, Study Director — Jilin University 1st Hospital Cardiovascular Center
Locations (1):
- Jilin University 1st Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided
When the investigation is completed,we will share it with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Derivation Cohort: Patients enrolled in the study in Jilin University First Hospital, no interventions will be administrated
- Validation Cohort: Patiens enrolled in the study in First affiliated Hospital of Shantou University, no interventions will be administrated
Period: Overall Study
Arm/Group | Derivation Cohort | Validation Cohort
Started | 6038 | 2438
Completed | 5185 | 2058
Not Completed | 853 | 380

BASELINE CHARACTERISTICS:
Population: A total of 5185 patients (average age 59.85 ± 9.95 years, 68.60% male) from the derivation cohort and 2058 patients (average age 60.00 ± 10.22 years, 68.71% male) from the validation cohort were included in the analysis, respectively.
Groups:
- Derivation Cohort: Patients enrolled in Jilin University First Hospital, no interventions will be administrated
- Validation Cohort: Patients enrolled in First Affiliated Hosptal of Shantou University, no interventions will be administrated
- Total: Total of all reporting groups
Arm/Group | Derivation Cohort | Validation Cohort | Total
Number analyzed (Participants) | 5185 | 2058 | 7243
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.846 (9.95) | 60.00 (10.22) | 59.96 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1628 | 644 | 2272
  Male | 3557 | 1414 | 4971
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History or Diabetes Mellitus [Number; unit: participants] | 1329 | 550 | 1879
Hypertension [Count of Participants; unit: Participants] | 2721 | 1073 | 3794
Dyslipidaemia [Count of Participants; unit: Participants] | 1640 | 515 | 2155
Current smoker [Count of Participants; unit: Participants] | 2914 | 1202 | 4116
History of drinking [Count of Participants; unit: Participants] | 764 | 327 | 1091
History of stroke/TIA [Count of Participants; unit: Participants] | 379 | 170 | 549
History of PVD [Count of Participants; unit: Participants] | 88 | 42 | 130
History of heart failure [Count of Participants; unit: Participants] | 137 | 58 | 195
Previous CABG [Count of Participants; unit: Participants] | 144 | 65 | 209
Previous PCI [Count of Participants; unit: Participants] | 104 | 46 | 150
Previous MI [Count of Participants; unit: Participants] | 357 | 114 | 471
AMI as admitting diagnosis [Count of Participants; unit: Participants] | 3160 | 1258 | 4418
Cardiogenic shock [Count of Participants; unit: Participants] | 113 | 17 | 130

OUTCOME MEASURES:

1. Primary Outcome: Very Late Stent Thrombosis
Description: very late stent thrombosis demonstrated by coronary angiography
Time Frame: Five years
Measure: Count of Participants; unit: Participants
Arm/Group | Derivation Cohort | Validation Cohort
Number analyzed (Participants) | 5185 | 2058
Participants | 92 | 35

ADVERSE EVENTS:
Time Frame: five years
Arm/Group | Derivation Cohort | Validation Cohort
All-Cause Mortality (participants affected / at risk) | 316/6038 | 132/2438
Serious Adverse Events (participants affected / at risk) | 0/6038 | 0/2438
Other Adverse Events (participants affected / at risk) | 0/6038 | 0/2438

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less